CLINICAL TRIAL: NCT02666768
Title: Open-label Early Phase 2 Study With a Single Arm of Interferon Gamma-1b Treatment of Osteopetrosis
Brief Title: ACTIMMUNE in Intermediate Osteopetrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: University of Minnesota (Other); Horizon Pharma Ireland, Ltd., Dublin Ireland (Industry)
Responsible Party: Principal Investigator, Lynda E Polgreen, Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21549-01
Record Dates: First submitted 2015-06-23; First posted 2016-01-28 (Estimated); Results first posted 2023-10-11 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Osteopetrosis
MeSH Terms: conditions — Osteopetrosis | interventions — interferon gamma-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gamma interferon-1b (Experimental): Gamma interferon-1b 100 mcg subcutaneous (SC) 3 times weekly for 12 months
  Interventions: Drug: Interferon gamma-1b

INTERVENTIONS:
Drug: Interferon gamma-1b — gamma interferon-1b dose escalation over first 4 weeks of study to 100 mcg SC 3 times weekly
  Other Names: ACTIMMUNE

SUMMARY:
This study evaluates the effects of ACTIMMUNE (IFN-γ1b) in children and adults with intermediate osteoporosis. All participants will receive treatment with ACTIMMUNE for 12 months. The investigators hypothesize that ACTIMMUNE will be tolerated by participants for the full 12 months and result in decreased disease severity.

DETAILED DESCRIPTION:
Osteopetrosis is a rare inherited metabolic bone disease characterized by impaired osteoclast function resulting in defective bone resorption and generalized high bone mass and mineral density (BMD). In patients with severe disease, this high bone mass compromises bone marrow space leading to marrow failure and frequent infections, along with hepatosplenomegaly from extramedullary hematopoiesis. Currently, the only treatment for individuals with severe forms of osteopetrosis is hematopoietic cell transplantation (HCT), however survival in patients with osteopetrosis treated with HCT is only around 55%. Therefore, this treatment is only indicated in select individuals with life-threatening complications of their disease. Thus additional treatments for osteopetrosis are needed both for individuals who are not candidates for HCT and to prolong the time until HCT is needed.

Interferon gamma (IFN-γ) is a naturally occurring cytokine that has been shown to have anti-microbial and anti-viral immunomodulatory effects, and is a potent stimulator of superoxide anion production which in turn promotes the formation and activation of osteoclasts. Two previous studies of IFN-γ1b in a small group of individuals with osteopetrosis found a decrease in trabecular bone area, an increase in marrow space, a decrease in the number of severe infections requiring antibiotic therapy, and an increase in superoxide generation by granulocyte-macrophage colonies.

Therefore, the investigators will conduct an early phase 2, multi-center, open-label, 12-month clinical trial of ACTIMMUNE (IFN-γ1b) treatment of patients with intermediate osteopetrosis to determine the following:

1. The feasibility and tolerability of interferon gamma-1b treatment for 1 year in patients with intermediate osteopetrosis. Specifically, i) the ability to enroll patients, and ii) continued treatment throughout the 1-year observational period.
2. Change in immunologic and hematologic function, bone mineral density and osteoclast function, physical function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of osteopetrosis; and
* Anemia (Hemoglobin <12 g/dL) not related to iron deficiency, or
* Neutropenia (Neutrophil count <1000 neutrophils/ul unsupported with cytokines), or
* Thrombocytopenia (Platelet count <50,000 cells x 109/L), or
* History of impaired bone healing, or
* ≥ 1 serious infection over prior year defined as requiring hospitalization and/or IV antibiotics, and
* Age > 1 year; and
* Ability to travel to a study center for every 3-6 month study visits; and
* Patient or parent/legal guardian is able and willing to provide informed consent. For patients 7 to 17 years of age, assent must also be provided.

Exclusion Criteria:

* 12 months or fewer following HCT;
* Pregnancy or breastfeeding;
* Known or suspected allergy to interferon gamma-1b or related products;
* Participation in simultaneous therapeutic study that involves an investigational study drug or agent within 4 weeks of study enrollment;
* ALT greater than 3 fold higher than normal; or
* Any other social or medical condition that the Investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated or be detrimental to the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda E Polgreen, MD, MS, Principal Investigator — Los Angeles BioMedical Research Center at Harbor-UCLA
Locations (2):
- United States (2):
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Minnesota, Minneapolis, Minnesota

REFERENCES:
- [Derived] Lertwilaiwittaya P, Suktitipat B, Khongthon P, Pongsapich W, Limwongse C, Pithukpakorn M. Identification of novel mutation in RANKL by whole-exome sequencing in a Thai family with osteopetrosis; a case report and review of RANKL osteopetrosis. Mol Genet Genomic Med. 2021 Jul;9(7):e1727. doi: 10.1002/mgg3.1727. Epub 2021 May 30. PMID 34056870

RESULTS

PARTICIPANT FLOW:
Groups:
- Gamma Interferon-1b: Gamma interferon-1b 100 micrograms (mcg) subcutaneously (SC) 3 times weekly for 12 months
  Interferon gamma-1b: gamma interferon-1b dose escalation over first 4 weeks of study to 100 mcg SC 3 times weekly
Period: Overall Study
Arm/Group | Gamma Interferon-1b
Started | 5
Completed | 1
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Gamma Interferon-1b
Number analyzed (Participants) | 5
Age, Continuous [Median (Full Range); unit: years] | 36.9 [15.1 to 59.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Genotype [Count of Participants; unit: Participants] — Genetic testing done as part of routine clinical care was collected when available. When not available this outcome was defined as "Unknown".
  Participants
    Chloride Voltage-Gated Channel 7 (CLCN7) mutation | 3
    T cell immune regulator 1 (TCIRG) mutation | 1
    Unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Related Adverse Events CTCAE v4.0 Grade 3 or Higher
Description: Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 defines a Grade 4 event as having life-threatening consequences, and/or urgent intervention indicated.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Gamma Interferon-1b: Gamma interferon-1b 100 mcg SC 3 times weekly for 12 months
  Interferon gamma-1b: gamma interferon-1b dose escalation over first 4 weeks of study to 100 mcg SC 3 times weekly
Arm/Group | Gamma Interferon-1b
Number analyzed (Participants) | 5
Participants | 0

2. Secondary Outcome: Percent Change From Baseline in Bone Mineral Density (BMD)
Description: BMD measured by peripheral quantitative computed tomography (pQCT) in bone area w/ BMD<169mg/m3
Time Frame: 6 months
Population: 1 participants withdrew due to flu-like side effects prior to 2nd pQCT measurement.
  1 participant has no data for this measurement due to size of pQCT gantry.
Measure: Median (Full Range); unit: percent change
Arm/Group | Gamma Interferon-1b
Number analyzed (Participants) | 3
percent change | 0 [-15 to 2]

3. Secondary Outcome: Change From Baseline in White Blood Cell Count (WBC)
Time Frame: 6 months
Population: Only 1 participant completed study to 12 months, so 6 month data are reported here.
Measure: Median (Full Range); unit: x1000 cells/uL
Arm/Group | Gamma Interferon-1b
Number analyzed (Participants) | 4
x1000 cells/uL | -0.5 [-1.2 to 1]

4. Secondary Outcome: Change From Baseline in Pain
Description: Survey name: RAND 36-Item Health Survey (Version 1.0) Scale name: Pain Scale range: 0-100; Higher score means less pain
Time Frame: 6 months
Population: One participant was <18 years old so did not complete the RAND 36-Item Health Survey
Measure: Least Squares Mean (95% Confidence Interval); unit: change in units on the pain scale
Arm/Group | Gamma Interferon-1b
Number analyzed (Participants) | 4
change in units on the pain scale | -0.8 [-2.0 to 0.3]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from day 1 to end of study or participant withdrawal, up to year 1.
Arm/Group | Gamma Interferon-1b
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gamma Interferon-1b (N=5)
Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Hyperglycemia (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 4 (5)
Flu-like reaction (General disorders) | 5 (13)
Injection site reactions (General disorders) | 3 (11)
Sinusitis/sinus pain/sinus congestion (Infections and infestations) | 2 (4)
Bone pain - generalized (Musculoskeletal and connective tissue disorders) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (5)
Headache (Nervous system disorders) | 4 (8)
Proteinuria (Renal and urinary disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations of this study include the small sample size, heterogeneity of the population, and difficulty obtaining endpoint measurements due to high withdrawal rate, all resulting in limited data for interpretation. Despite these limitations, this study provides information on the longest follow-up of treatment with interferon gamma-1b in this population and identified an approach to make the treatment tolerable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT02666768/Prot_SAP_000.pdf